CLINICAL TRIAL: NCT04470362
Title: Beni-Suef University
Brief Title: Effect of Proprioceptive Training on Muscle Fatigue in Older Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ayman Mohamed (Other)
Responsible Party: Sponsor-Investigator, Ayman Mohamed, Beni-Suef University, Beni-Suef University
Organization: Beni-Suef University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 250982
Record Dates: First submitted 2020-07-10; First posted 2020-07-14 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Proprioceptive Disorders
MeSH Terms: conditions — Somatosensory Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (Placebo Comparator): The control group will receive an isokinetic strengthening program for the quadriceps muscles. Twenty-four strengthening session will be performed using an isokinetic device. The exercise program begins with 60% of the mean peak torque, and the patient reaches this intensity by auditory biofeedback. An increasing dose program will be used in the first 5 sessions (1 set to 5 sets), and a dose of 6 sets will be applied from the sixth to twenty-fourth sessions, with the density rising from 60% to 80% of the mean peak torque according to the patient tolerance. Each set consisted of 5 repetitions of concentric (Con/Ecc) contraction in angular velocities of 30°/second and 120°/second for extensors. This program accomplished significant results in increasing quadriceps power and strength.
  Interventions: Device: Isokinetic dynamometer
- Study group (Experimental): * Participants in the study group will perform the same exercise parameters used in the control group but in a different manner.
  * The isokinetic exercise will be done with a closed eye to improve the proprioception function. This exercise will be performed for 6 sets.
  * Additional training will be performed by the application of three vibrators above and on both sides of the knee joint to improve the function of the Pacinian and Meissner corpuscles which is one of the included receptors in the sensation of the fatigue.
  Interventions: Device: Isokinetic dynamometer

INTERVENTIONS:
Device: Isokinetic dynamometer — an isokinetic strengthening program for the quadriceps muscles. Twenty-four strengthening session will be performed using an isokinetic device. The exercise program begins with 60% of the mean peak torque, and the patient reaches this intensity by auditory biofeedback. An increasing dose program will be used in the first 5 sessions (1 set to 5 sets), and a dose of 6 sets will be applied from the sixth to twenty-fourth sessions, with the density rising from 60% to 80% of the mean peak torque according to the patient tolerance. Each set consisted of 5 repetitions of concentric (Con/Ecc) contraction in angular velocities of 30°/second and 120°/second for extensors. This program accomplished significant results in increasing the quadriceps power and strength.

SUMMARY:
Summary Muscle fatigue is a serious problem commonly occur in older ages. Muscle fatigue disturbs both daily life activities and rehabilitation tolerance in elderlies. Muscle fatigue happens due to the motor or sensory dysfunctions. The previous interventions focused mainly on the motor causes of muscle fatigue, however the important role of the sensory system in driving the motor system. It has been demonstrated that proprioceptors are mainly responsible for sensing the muscle fatigue. Objectives: This study will be conducted to investigate 1. The effect of proprioception training on reducing the occurrence of muscle fatigue in elderlies. 2. The effect of proprioceptive training on delaying the deterioration in electromyographical data from muscles of lower limbs.

DETAILED DESCRIPTION:
Study protocol A single blinded randomized parallel study design will be used in this study. 40 participants will be recruited for this study aged from 65 to 90 years old. The randomization will be performed using simple envelop methods. Participants will be divided into two groups, control and study groups. The control group will receive an isokinetic strengthening program for the quadriceps muscles. Twenty-four strengthening session will be performed using an isokinetic device. The exercise program begins with 60% of the mean peak torque, and the patient reaches this intensity by auditory biofeedback. An increasing dose program will be used in the first 5 sessions (1 set to 5 sets), and a dose of 6 sets will be applied from the sixth to twenty-fourth sessions, with the density rising from 60% to 80% of the mean peak torque according to the patient tolerance. Each set consisted of 5 repetitions of concentric (Con/Ecc) contraction in angular velocities of 30°/second and 120°/second for extensors. This program accomplished significant results in increasing the quadriceps power and strength.

Participants in the study group will perform the same exercise parameters used in the control group but in a different manner. The isokinetic exercise will be done with a closed eye to improve the proprioception function. This exercise will be performed for 6 sets. We will add another set, in which the participant will be instructed that the range of motion of the knee joint will be divided into three ranges, the outer range (from 0 to 90 degrees of knee flexion), the middle range (90 degrees of flexion) and inner range (from 90 degrees to 145 degree of flexion). During this set, the isokinetic device will be stopped at a different joint angle and the participant will be asked to identify at which range the knee joint is in. This modification is directed to improve the function of muscle spindles and Golgi tendon organs.

Additional training will be performed by the application of three vibrators above and on both sides of the knee joint to improve the function of the Pacinian and Meissner corpuscles which is one of the included receptors in the sensation of the fatigue. This vibration will be set at a subsensory intensity (Stochastic theory39) and a frequency fluctuating frequency from 50 Hz to 250 Hz to train both receptors40 and it will be performed for 20 min/each session. This programs will be performed for three sessions/week for two months.

The primary outcomes measure will be the electromyographical analysis of quadriceps muscle at the onset of muscle fatigue and after recovery. The secondary outcome measures will include the Fatigue Index (FI) and the Rating-of-Fatigue Scale. These measurements at baseline, After one month, After two months.

ELIGIBILITY:
Inclusion Criteria:

* Elderlies over 65 years old

Exclusion Criteria:

* No previous history of lower extremity trauma, serious metabolic, neurological, muscular, inflammatory or cardiovascular diseases

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-04-01 (Estimated); Primary Completion 2021-04-01 (Estimated); Study Completion 2021-09-01 (Estimated)

PRIMARY OUTCOMES:
EMG of quadriceps muscles | Two Months
  The electromyographical analysis of quadriceps muscle at the onset of muscle fatigue and after recovery

SECONDARY OUTCOMES:
The fatigue index (FI) | Two months
  The fatigue index (FI) was calculated according to the following formula (Bar-Or, 1987): FI = (maximal pedal speed - minimal pedal speed) / maximal pedal speed * 100.
Rating-of-Fatigue Scale | Two months
  he ROF scale consists of 11 numerical points that range from 0 to 10. There are also five descriptors and five diagrams to help the person understand the scale and make a rating.
  The Rating of fatigue scale consists of 11 numerical points that range from 0 to 10. There are also five descriptors and five diagrams to help the person understand the scale and make a rating.

CONTACTS AND LOCATIONS:
Locations (1):
- Beni Suef University, Banī Suwayf, Beni Suweif Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided